CLINICAL TRIAL: NCT02825745
Title: A Feasibility Study of the Use of Betashot, a Medium Chain Triglyceride- Based (MCT) Food for Special Medical Purposes (FSMP) in Children and Adults With Epilepsy.
Brief Title: Use of Betashot in Children and Adults With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCT-BETS-14082015-01; 181054 (Other: IRAS)
Record Dates: First submitted 2015-09-07; First posted 2016-07-07 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Nervous System Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Betashot (Other): Children:will take Betashot as a proportion of their daily energy requirements calculated from the dietary information obtained during Visit A for up to 12 weeks.
  Adults:will introduce Betashot and increase the amount taken in ml incrementally for up to 12 weeks.
  Interventions: Dietary Supplement: Betashot

INTERVENTIONS:
Dietary Supplement: Betashot — Betashot is a Food for Special Medical Purposes (FSMP). Suitable for use from 3 years of age.
  Other Names: MCT based emulsion

SUMMARY:
In brief, this research is a prospective, feasibility study to evaluate the use of Betashot- a medium chain triglyceride- based (MCT) food for special medical purposes (FSMP) in children and adults diagnosed with epilepsy.

MCT is a type of dietary fat used in the ketogenic diet.

DETAILED DESCRIPTION:
This study aims to explore the use of Betashot in a group of children and adults with epilepsy who are consuming their normal diets, but limiting intakes of foods high in carbohydrate and sugars.

The participants will be required to drink Betashot to enable the following assessment:

1. Tolerance (side effects such as bloating or cramps)
2. Acceptability (flavour, texture, taste)
3. Compliance (how easy it is to use Betashot at the advised quantity, as part of their daily diet)

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3-18 years with symptoms of epilepsy continuing despite adequate levels of anti-epileptic medication, either with a diagnosis of Dravet syndrome or another early onset epilepsy, the result of a genetic mutation.

   Adults (aged over 18) with symptoms of epilepsy continuing despite adequate levels of anti-epileptic medication.
2. Participant/Parent/guardian to comply with the study protocol and participate in active monitoring of tolerance, acceptability and compliance of Betashot via a written record, and to complete questionnaires.

Exclusion Criteria:

1. Children < 3 years of age
2. Children and adults free from epilepsy for > 4 weeks
3. Medical conditions that contra-indicate the use of MCT
4. Inability to comply with the study protocol.
5. Currently on a ketogenic diet
6. Children and adults who are totally enterally fed.
7. Females who are pregnant or planning to become pregnant during the study.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Palatability | 12 weeks
  The primary outcome measure for the study is to determine, via a questionnaire, the palatability of Betashot
Gastrointestinal tolerance | 12 weeks
  The primary outcome measure for the study is to determine, via a questionnaire, the GI tolerance of Betashot
Compliance | 12 weeks
  The primary outcome measure for the study is to determine, via a questionnaire, the patient compliance with Betashot

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Walker, Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No